CLINICAL TRIAL: NCT00393224
Title: Defining Markers of Susceptibility to Nasopharyngeal Carcinoma (NPC) Within High-Risk, Multiplex NPC Families
Brief Title: Defining the Clinical Utility of EBV Antibody Screening to Identify Individuals Susceptible to Nasopharyngeal Carcinoma (NPC) Within High-Risk, Multiplex NPC Families
Status: Terminated | Type: Observational
Why Stopped: Determined not to be human subject reseach
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905187; 05-C-N187; NCT00898248 (obsolete NCT alias)
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: Epidemiology; Nasopharyngeal Carcinoma; Genetic; Viruses; Cancer; NPC
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Nasopharyngeal Carcinoma; Virus Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort: hospital based family cohort

SUMMARY:
In an effort to identify genetic factors linked to the development of nasopharyngeal cancer (NPC), the researchers identified and sampled 2,394 individuals from Taiwanese families in which two or more relatives had been diagnosed with NPC. Serum from these individuals was tested for three anti-Epstein-Barr virus (EPV) antibodies associated with elevated risk of NPC. Results indicate that apparently healthy individuals from high-risk families have a nearly threefold elevation in their EBV antibody prevalence compared with the general population. However, the clinical implications of this finding are not yet understood.

To clarify the implications, the 2,394 unaffected individuals from the multiplex family study will be invited to participate in the current study. Approximately 1,600 individuals are expected to participate.

Participants will have an ear, nose, and throat examination to determine if they have occult or symptomatic NPC. Their levels of EBV antibody at the time of initial recruitment will be correlated with NPC detection in the period between initial recruitment and the present study. Participants will also be asked to complete a brief risk factor questionnaire and to donate blood, saliva, a nasopharyngeal swab, nasopharyngeal tissue, and urine for future studies.

Currently, no accepted clinical management protocol exists for screening unaffected members from families at high risk of NPC development. Results from this study have the potential to significantly impact the clinical management and follow-up of individuals with a family history of NPC.

DETAILED DESCRIPTION:
The purpose of this proposed study is to evaluate the clinical utility of serum EBV antibody testing for the identification of individuals at increased risk of nasopharyngeal carcinoma (NPC) within high-risk, NPC multiplex families.

2,394 unaffected individuals from Taiwanese families, in which two or more relatives have been diagnosed with NPC, have been identified and sampled as part of an ongoing collaboration to identify genetic factors linked to NPC development. Serum from these individuals has been tested for three anti-EBV antibodies (VCA IgA, EBNA1 IgA, and anti-DNase) known to be associated with elevated risk of prevalent and incident NPC in general population studies. Results from testing of our study population indicate that apparently healthy individuals from high-risk multiplex families have a near 3-fold elevation in their EBV antibody prevalence when compared to the EBV antibody prevalence observed in the general community for these same EBV markers. However, the clinical implications of this apparent elevation in EBV antibody reactivity are not yet understood.

Therefore, we propose to evaluate whether individuals within our previously conducted high-risk family study with elevations in EBV antibody levels are at increased risk of incident NPC. Individual markers (VCA IgA, EBNIA1 IgA and anti-DNase antibodies) and combinations of markers will be evaluated to determine their performance as screening tests for NPC risk in high-risk multiplex families.

To achieve this goal, we propose to invite the 2,394 unaffected individuals from our multiplex family study, defined as those families with greater than or equal to 2 NPC. As a result of our recruitment efforts, we expect approximately 1,600 subjects to participate in an ear, nose, and throat (ENT) examination by an expert otolaryngologist to determine whether any of these individuals has occult or symptomatic NPC. We will correlate the three EBV antibody screening tests performed at the time of initial recruitment into our family study with NPC detection in the period between initial recruitment into the family study and the present study (median time between original EBV antibody testing and clinical evaluation = 5.5 years; range = less than 1 year - 10 years).

In addition to histopathological specimens collected for NPC diagnosis, participants in this study will be asked to agree to a brief risk factor questionnaire and to donate blood, saliva, a nasopharyngeal swab, nasopharyngeal tissue, and urine for future studies.

No accepted clinical management protocol exists for screening unaffected members from families at high-risk of NPC development. Results from this study have the potential to significantly impact the clinical management and follow-up of individuals with a family history of NPC.

ELIGIBILITY:
* INCLUSION CRITERIA:

The 2,394 unaffected family members who previously participated in the family study of nasopharyngeal carcinoma (NPC) in Taiwan between 1996 and 2004.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a hospital based family cohort
Sampling Method: Non-Probability Sample
Enrollment: 952 (Actual)
Dates: Start 2005-07-05 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
NPC | ongoing
  NPC

CONTACTS AND LOCATIONS:
Overall Officials: Allan Hildesheim, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Taiwan University, Taiwan, China

REFERENCES:
- [Background] Cohen JI. Epstein-Barr virus infection. N Engl J Med. 2000 Aug 17;343(7):481-92. doi: 10.1056/NEJM200008173430707. No abstract available. PMID 10944566
- [Background] Hsu JL, Glaser SL. Epstein-barr virus-associated malignancies: epidemiologic patterns and etiologic implications. Crit Rev Oncol Hematol. 2000 Apr;34(1):27-53. doi: 10.1016/s1040-8428(00)00046-9. PMID 10781747
- [Background] Zeng Y, Zhang LG, Wu YC, Huang YS, Huang NQ, Li JY, Wang YB, Jiang MK, Fang Z, Meng NN. Prospective studies on nasopharyngeal carcinoma in Epstein-Barr virus IgA/VCA antibody-positive persons in Wuzhou City, China. Int J Cancer. 1985 Nov 15;36(5):545-7. doi: 10.1002/ijc.2910360505. PMID 4055129